CLINICAL TRIAL: NCT03673072
Title: Neoadjuvant Chemotherapy With Gemcitabine Plus Cisplatin Followed by Radical Liver Resection Versus Immediate Radical Liver Resection Alone With or Without Adjuvant Chemotherapy in Incidentally Detected Gallbladder Carcinoma After Simple Cholecystectomy or in Front of Radical Resection of BTC (ICC/ECC) - A Phase III Study of the German Registry of Incidental Gallbladder Carcinoma Platform (GR) - The AIO/ CALGP/ ACO- GAIN-Trial -
Brief Title: Neoadjuvant Chemotherapy With Gemcitabine Plus Cisplatin Followed by Radical Liver Resection Versus Immediate Radical Liver Resection Alone With or Without Adjuvant Chemotherapy in Incidentally Detected Gallbladder Carcinoma After Simple Cholecystectomy or in Front of Radical Resection of BTC
Acronym: GAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAIN/GEM/CIS; 2017-004444-38 (EudraCT Number); AIO-HEP-0118/ass (Other: AIO)
Record Dates: First submitted 2018-09-03; First posted 2018-09-17 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Incidental Gallbladder Carcinoma; Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (gemcitabine plus cisplatin) (Experimental): Patients assigned to arm A will receive treatment with gemcitabine plus cisplatin. Chemotherapy will be administered for 3 cycles preoperatively (neoadjuvant part) and for 3 cycles postoperatively (adjuvant part).
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Procedure: Oncologically radical margin-free (R0) resection
- Arm B (standard postoperative management) (Active Comparator): Patients assigned to arm B will receive surgery directly, without receiving perioperative chemotherapy (Standard of Care / SOC). After surgery, adjuvant chemotherapy can be administered by investigator's choice.
  Interventions: Procedure: Oncologically radical margin-free (R0) resection; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine (1000 mg/m2) in 250-500 ml 0.9% saline every three weeks on days 1 and 8 intravenously
  Arms: Arm A (gemcitabine plus cisplatin)
Drug: Cisplatin — Cisplatin (25 mg/m2) every three weeks on days 1 and 8 intravenously, in 1000 ml 0.9% saline with KCl 20 mmol and MgSO4 8 mmol during the one hour cisplatin infusion followed by 500 ml 0.9% saline over 30 minutes prior to gemcitabine; with adequate pre- and posthydration
  Arms: Arm A (gemcitabine plus cisplatin)
Procedure: Oncologically radical margin-free (R0) resection — Oncologically radical margin-free (R0) resection
Drug: Adjuvant chemotherapy — Can be selected by Investigator's Choice
  Arms: Arm B (standard postoperative management)

SUMMARY:
Neoadjuvant chemotherapy with gemcitabine plus cisplatin followed by radical liver resection versus immediate radical liver resection alone with or without adjuvant chemotherapy in incidentally detected gallbladder carcinoma after simple cholecystectomy or in front of radical resection of BTC (ICC/ECC)

DETAILED DESCRIPTION:
The aim of the study is to investigate whether induction chemotherapy followed by radical re-resection (and - if possible - postoperative chemotherapy) in incidental gallbladder carcinoma (IGBC) or in front radical resection in biliary tract cancer (BTC) (intrahepatic cholangiocarcinoma (ICC)/ extrahepatic cholangiocarcinoma (ECC)) prolongs overall survival without impaired quality of life compared to immediate radical surgery alone with or without adjuvant chemotherapy (investigator's choice) in patients with IGBC, or BTC (ICC/ECC). One of the most important secondary objectives is to raise awareness for the necessity of a radical second surgery as well as to improve the adherence to the treatment guidelines in IGBC. Further secondary objectives are safety and tolerability of the treatment as well as quality of life.

ELIGIBILITY:
Inclusion criteria

1. Incidental gallbladder carcinoma (IGBC), gallbladder carcinoma (GBC) () or Biliary tract cancer (BTC) (intrahepatic, hilar or distal Cholangiocarcinoma (CCA)) scheduled for complete resection (mixed tumor entities with hepatocellular carcinoma are excluded).
2. No prior partial or complete tumor resection for BTC (intrahepatic, hilar or distal CCA), and for IGBC/GBC prior Cholecystectomy is allowed.
3. Exclusion of distant metastases by CT or MRI of abdomen, pelvis, and thorax, bone scan or MRI (if bone metastases are suspected due to clinical signs). Exclusion of the infiltration of any adjacent organs or structures by CT or MRI, indicating an unresectable situation.
4. ECOG performance status of 0, 1, or 2.
5. Estimated life expectancy > 3 months.
6. Female and male patients1 ≥18 years.
7. Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures
8. No previous or preceding cytotoxic or targeted therapy for BTC or IGBC/GBC.
9. No previous malignancy within two years or concomitant malignancy, except for curatively treated basal cell carcinoma of the skin, in situ carcinoma of the cervix, and prostate cancer
10. No severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction in the last three months, significant arrhythmia).
11. Absence of psychiatric disorder precluding understanding of information of trial related topics and giving informed consent.
12. No serious underlying medical conditions (judged by the investigator), that could impair the ability of the patient to participate in the trial.
13. A) Females of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 7 months after the last study treatment.

    A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (has not had ≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

    B) Males must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agree to refrain from donating sperm, as defined below:

    With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of 1% per year during the treatment period and for at least 6 months after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period. Men with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy.
14. No pregnancy or lactation.
15. Adequate hematologic function: ANC ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 9 g/dl or ≥ 5.59 mmol/L; prior transfusions for patients with low hemoglobin are allowed
16. Adequate liver function as measured by serum transaminases (AST and ALT) ≤ 5 x ULN and bilirubin ≤ 3 x ULN.
17. Adequate renal function, i.e. serum creatinine ≤ 1.5 x institutional ULN, a calculated glomerular filtration rate ≥ 30 mL/min.
18. Adequate coagulation functions as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients receiving warfarin/ phenprocoumon must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to randomization.
19. No active uncontrolled infection, except chronic viral hepatitis under antiviral therapy (patients on long-term antibiotics are eligible provided signs of active infection have been resolved).
20. No concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days or five half-lives (whichever is longer) prior to randomization.
21. Negative serum pregnancy test within 7 days of starting study treatment in pre-menopausal women and women <1 year after the onset of menopause Please note that after randomization for patients in Arm A the histological confirmation of BTC or GBC must be performed before administering chemotherapy. For IGBC histological confirmation should already have been performed.

For Arm B patients the histological confirmation can be performed after surgery with material from the surgery.

Exclusion criteria

1. Known hypersensitivity against gemcitabine or cisplatin
2. Other known contraindications to gemcitabine or cisplatin
3. Clinically significant valvular defect
4. Past or current history of other malignancies not curatively treated and without evidence of disease for more than two years, except for curatively treated basal cell carcinoma of the skin, in situ carcinoma of the cervix, and prostate cancer
5. Locally unresectable tumor or metastatic disease:

   * Radiological evidence suggesting inability to resect with curative intent whilst maintaining adequate vascular inflow and outflow, and sufficient future liver remnant
   * Radiological evidence of direct invasion into adjacent organs
   * Radiological evidence of extrahepatic metastatic disease
6. Other severe internal disease or acute infection
7. Chronic inflammatory bowel disease
8. Receiving chronic antiplatelet therapy, including aspirin (Once-daily aspirin use (maximum dose 325 mg/day) is permitted), nonsteroidal anti-inflammatory drugs (including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents.
9. History of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during 3 months prior to randomization.
10. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or ascites.
11. On-treatment participation in another clinical study 30 days or five half-lives (whichever is longer) prior to inclusion and during the study
12. Pregnant or breast feeding patient, or patient is planning to become pregnant within 7 months after the end of treatment.
13. Patients in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4)
14. Any other concurrent antineoplastic treatment including irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint is overall survival (OS) | up to 6 years follow-up

SECONDARY OUTCOMES:
Quality of life (EORTC QLQ-C30) | every 3 weeks until EOT andt then every 3 months up to 6 years of follow-up
  "European Organisation for the Research and Treatment of Cancer" Quality of Life Questionnaire Core 30. The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients.
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
PFS (Progression free surviva) rates at 3 and 5 years | at 3 and 5 years after randomization
OS (overall survival) rates at 3 and 5 years | at 3 and 5 years after randomization
Progression free survival (PFS) | up to 6 years after randomization
R0- resection rate | 2 weeks after surgery (Arm A: 14 weeks after randomization; Arm B: 2 weeks after randomization)
Toxicity, graded using CTC adverse events criteria version CTCAE V 5.0 | up to 6 years after randomization
Number of patients with any serious perioperative morbidity or mortality | up to 30 and 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten O Goetze, PD Dr., Principal Investigator — Krankenhaus Nordwest
Locations (1):
- Krankenhaus Nordwest gGmbH, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Goetze TO, Bechstein WO, Bankstahl US, Keck T, Konigsrainer A, Lang SA, Pauligk C, Piso P, Vogel A, Al-Batran SE. Neoadjuvant chemotherapy with gemcitabine plus cisplatin followed by radical liver resection versus immediate radical liver resection alone with or without adjuvant chemotherapy in incidentally detected gallbladder carcinoma after simple cholecystectomy or in front of radical resection of BTC (ICC/ECC) - a phase III study of the German registry of incidental gallbladder carcinoma platform (GR)- the AIO/ CALGP/ ACO- GAIN-trial. BMC Cancer. 2020 Feb 14;20(1):122. doi: 10.1186/s12885-020-6610-4. PMID 32059704